CLINICAL TRIAL: NCT01755000
Title: A Pilot Feasibility Study of Hypotensive Hematopoietic Malignancy Patients' USCOM Readings
Brief Title: Study of Hypotensive Hematopoietic Malignancy Patients' USCOM Readings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201206070
Record Dates: First submitted 2012-12-18; First posted 2012-12-21 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: Leukemia; Lymphoma; Paraproteinemias; Multiple Myeloma; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia; Lymphoma; Paraproteinemias; Multiple Myeloma; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aim 1: Hemodynamically Healthy Patients (Other): Nurse 1 will perform an USCOM scan and record values of Vpk and SV on the clinical data sheet.
  Nurse 2 will perform the USCOM second scan within five minutes of Nurse 1's scan and record the values of Vpk and SV on the clinical data sheet.
  Nurse 1 and 2 will be blinded to each other's scans by using separate clinical data forms
  Interventions: Procedure: USCOM scan
- Aim 2: Hemodynamically Unstable Patients (Other): Nurse 1 will perform an USCOM scan and record values of Vpk and SV on the clinical data sheet.
  Nurse 2 will also be notified of the hypotensive event, will then perform the USCOM second scan within five minutes of PI's scan and record the values of Vpk and SV on the clinical data sheet.
  The two USCOM scans will be completed within 10 minutes of the hypotensive episode.
  Nurse 1 and Nurse 2 will be blinded to each other's scans by using separate clinical data forms.
  Interventions: Procedure: USCOM scan
- Aim 3: Hemodynamically Unstable Patients + Fluid Bolus (Other): At the time that an enrolled patient meets one of the following criteria; SBP drops below 95 mmHg or MAP drops below 65 mmHg the PI will be notified to PI to perform the USCOM scan and record the Vpk, SV, systolic blood pressure and mean arterial pressure on the clinical data sheet within 10 minutes of the hypotensive episode, prior to the patient receiving a fluid bolus (fluid bolus is part of standard of care).
  The USCOM scan will then be repeated within 5 minutes after fluid bolus delivery.
  Before the hemodynamically unstable patient receives subsequent fluid boluses (multiple boluses are common standard of care), the PI will perform an USCOM scan. Then within 5 minutes after the delivered fluid bolus, the PI will perform another USCOM scan. This will continue, until no further boluses are prescribed.
  Interventions: Procedure: USCOM scan; Procedure: Fluid Bolus

INTERVENTIONS:
Procedure: USCOM scan
Procedure: Fluid Bolus
  Arms: Aim 3: Hemodynamically Unstable Patients + Fluid Bolus

SUMMARY:
The purpose of this study is to test how practical it is to use the Ultrasonic Cardiac Output Monitor (USCOM), an FDA-approved device, on oncology patients (specifically those with blood cancers). Additionally, the researchers will learn if the USCOM gives additional information about patients' conditions when their blood pressures drop and they are treated with intravenous fluids.

ELIGIBILITY:
Inclusion Criteria:

-≥ 18 years of age

* English speaker
* Diagnosis of blood dyscrasia, hematopoietic malignancy, or condition that may requires HSCT

Exclusion Criteria:

* Obstruction of the suprasternal notch that prevents placing the USCOM probe in the correct location
* Tracheostomy or endotracheal tube that prevents placing USCOM probe in the correct location
* Inability to lie flat, on left or right side, or with the head of bed at a 30 degree angle for the USCOM exam (ex. due to respiratory distress or physiologic reasons)
* Impairment by a psychiatric, cognitive, or physiologic disorder that limits ability to understand explanation of study and give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2012-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
What is the inter-rater agreement between multiple independent USCOM users measuring stroke volume (SV) and peak velocity (Vpk) whose systolic blood pressures (SBPs) and mean arterial pressures (MAPs) are stable (SBP above 95 mmHg and MAP above 65 mmHg)? | 1 day (one time event for patient)
  Pairs of USCOM measurements from multiple raters for SV and Vpk, both of which are interval-level measures. Inter-rater reliability will be assessed using the Intraclass Correlation Coefficient (ICC); our design fits into case 1 using the Shrout and Fleiss (1979) classification system.
What is the inter-rater agreement between multiple independent USCOM users measuring SV and Vpk in hematopoietic malignancy patients whose SBPs drop below 95mmHg or MAPs drop below 65mmHg? | 1 day (one time event for patient)
  pairs of USCOM measurements from multiple raters for SV and Vpk. We will use the ICC to evaluate rater agreement here, as well, with the same sample size and the same confidence interval. For Aim 2, though, if the second rating cannot be completed within 5 minutes of the first, that episode will be excluded from the study.
In what percentage of patients is fluid bolus administration successful as measured by the current standard of care (MAP) and what is the level of agreement between the standard measure and USCOM readings in determining return to hemodynamic stability? | 1 day (one time event for patient)
  After two raters have measured SV and Vpk, bolus will be administered. Determining the success of bolus administration, we will simply record whether the clinician judged the bolus to be successful. In addition, one rater will measure SV and Vpk again using USCOM within 5 minutes of bolus administration. We will then calculate the percentage of patients whose stroke volume and peak velocity increased at least 15% after bolus administration using the post-bolus USCOM reading and the same rater's pre-bolus USCOM reading. We chose an increase of 15% based on a review of the research as the threshold that would best indicate a therapeutic response to bolus administration.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Parmentier, RN, BSN, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu